CLINICAL TRIAL: NCT03887637
Title: Real-world Effectiveness and Safety of Treatment With Direct Antiviral Agents (DAAs) in Patients With Chronic Hepatitis C and Cirrhosis in Southern Area of China
Brief Title: Real-world Effectiveness and Safety of Treatment With DAAs in Patients With CHC(Chronic Hepatitis C)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chaoshuang Lin, Professor/Chief physician, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: LinChaoShuang
Record Dates: First submitted 2019-03-15; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Danoprevir Sodium triple therapy: DNV(Danoprevir Sodium)/PegIFNα(Peginterferon α-2a)/RBV(Ribavirin) : (1) DNV : 100mg (one tablet) orally twice daily for 12 weeks. (2) PegIFNα: 180ug subcutaneous infection on abdomen or thigh once a week for 12 weeks. (3) RBV: 500mg (5 tablets) orally twice daily for 12 weeks in patients weighing less than 75kg; 600mg (6 tablets) orally twice daily for 12 weeks in patients weighing ≥75kg.
  Dosing time: In the morning, participants will be instructed to take DNV and RBV with food or one hour after food. The drugs are not allowed to be cut or divided. The interval between DNV and RBV dosing time should be 12±2 hours.
  Interventions: Drug: DAAs
- Sofosbuvir/ Velpatasvir therapy: Sofosbuvir/ Velpatasvir :500mg (two drugs in one tablet) orally once daily for 12 weeks.
  Interventions: Drug: DAAs
- Ombitasvir/Paritaprevir therapy: Ombitasvir/Paritaprevir: Ombitasvir two tablets orally once daily for 12 weeks; Paritaprevir one tablet orally twice daily for 12 weeks.
  Interventions: Drug: DAAs
- Grazoprevir/elbasvir therapy: Grazoprevir/elbasvir: 150mg (two drugs in one tablet) orally once daily for 12 weeks.
  Interventions: Drug: DAAs
- Daclatasvir/Asunaprevir therapy: Daclatasvir (60mg)one tablet once daily and Asunaprevir (100mg)one tablet twice daily for 24weeks
  Interventions: Drug: DAAs
- Danoprevir Sodium/Sofosbuvir therapy: Danoprevir Sodium: 100mg (one tablet) orally twice daily for 12 weeks;Sofosbuvir:400mg (one tablet) orally once daily for 12 weeks.
  Interventions: Drug: DAAs

INTERVENTIONS:
Drug: DAAs — Patients with CHC and cirrhosis who fulfills the indication of antiviral therapy will be administered with DAAs treatment.

SUMMARY:
This is a multi-center, open-label clinical study. This study was aimed to assess the real-world effectiveness and safety of treatment with listed DAAs in patients with CHC and cirrhosis in Southern area of China.

DETAILED DESCRIPTION:
This is a multi-center, open-label clinical study. This study was aimed to assess the real-world effectiveness and safety of treatment with listed DAAs in patients with CHC and cirrhosis in Southern area of China.

The primary objectives of this study is as follows:

To access the effectiveness and safety of 12-week/24-week treatment with listed DAAs in patients with CHC and cirrhosis in real-world clinical practice in Southern area of China. The proportion of participants with SVR12(Undetectable HCV RNA at 12 weeks after treatment completion RNA:Hepatitis C virus ribonucleic acid) was evaluated.

This study aims to enroll 30 patients with CHC and cirrhosis in each treatment group.

Patients with CHC and cirrhosis who fulfills the indication of antiviral therapy will be administered with DAAs treatment. After 12-week/2-week treatment, all the patients will be followed up for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with age >18 years old.
* HCV RNA ≥1×103IU/mL
* Genotype 1-6 HCV infection.
* Confirmed CHC defined as: (1)Confirmed HCV infection more than 6 months at baseline, including anti-HCV positive or HCV RNA positive for at least 6 months; (2)Confirmed HCV infection by liver biopsy one year before baseline.
* Negative pregnancy test for females of childbearing potential (18 years old to one year after menopause) at screening.
* Males and females of childbearing potential should agree to take mechanic contraceptives from screening to at least 6 months after discontinuation of treatment.
* Informed of, willing and able to comply with all of the protocol requirements and the investigational nature of the study.
* A signed written informed consent from patient.

Exclusion Criteria:

* History of clinically significant medical condition associated with other chronic liver disease (including hemochromatosis, autoimmune hepatitis, Wilson's disease, α1-antitrypsin deficiency, alcoholic liver disease, drug-induced liver injury).
* Stomach disorder that could interfere with the absorption of the study drug.
* Serious or active medical or psychiatric illness. If the participant has received more than 12 months of treatment and the condition is stable, or the participant does not need any medicine during the previous 12 months, the participant is allowed to enrollment.
* Uncontrolled serious cardiovascular disease (such as ventricular tachyarrhythmia, myocardial infarction, angina or coronary disease); or uncontrolled hypertension (systolic pressure ≥160mmHg and/or diastolic pressure ≥100mmHg); or clinically relevant ECG abnormalities.
* Serious respiratory or renal diseases.
* Serious hematological diseases or increased risk of anemia (such as Mediterranean anemia, sickle cell disease, spherocytosis, gastrointestinal bleeding).
* Uncontrolled diabetes or other endocrinological diseases.
* Suspension of malignant tumor.
* Participant who has received organ or bone-marrow allograft, or plans to receive organ transplantation during the treatment.
* Any confirmed significant allergic reactions against any drug, or the therapeutic drug and its metabolites.
* Uncontrolled autoimmune diseases, including but not limited to myositis, hepatitis, interstitial lung disease, interstitial nephritis, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, thyroiditis, psoriasis, rheumatoid arthritis, et al.
* Anti-HAV (IgM), anti-HEV (IgM) or anti-HIV positive. HBsAg-positive is not limited.
* Pregnancy or breast-feeding (non-breast-feeding is not included) female.
* History of drug and/or alcohol abuse within 6 months before screening that could interfere with evaluation.
* Participation in other clinical trial or an investigational drug 3 months before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects with age >18 years old
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-03-30 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
SVR(Sustained Virologic Response)12 | 12 weeks
  The proportion of participants with HCV RNA undetectable at 12weeks after treatment completion

SECONDARY OUTCOMES:
RVR (Rapid Virological Response)4 | 4 weeks
  The proportion of participants with HCV RNA undetectable at 4 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shuang C Lin, Professor, Principal Investigator — Third Sun Yat Sen

IPD SHARING:
Plan to Share IPD: Undecided